CLINICAL TRIAL: NCT05036538
Title: Decreasing Preoperative Stress to Prevent Postoperative Delirium and Postoperative Cognitive Decline in Cardiac Surgical Patients. A Randomized Controlled Trial on Relaxation Interventions Via Virtual Reality and Binaural Beats.
Brief Title: Decreasing Preoperative Stress to Prevent Postoperative Delirium and Postoperative Cognitive Decline in Cardiac Surgical Patients.
Acronym: DESTRESS-SURG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heart and Brain Research Group, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110/21
Record Dates: First submitted 2021-08-12; First posted 2021-09-05 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Preoperative Stress; Postoperative Cognitive Dysfunction; Postoperative Delirium
Keywords: Cardiac Surgery; Postoperative Cognitive Decline; Postoperative Delirium; Preoperative Stress; Relaxation Intervention; Virtual Reality; Binaural Beats
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — Methods; Smart Glasses

STUDY DESIGN:
Intervention Model Description: Randomized controlled intervention study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Surgeons, neurologists, and neuropsychologists who will be involved in the assessment of outcome variables will be blinded for randomization status. The intervention sessions will be conducted by a psychological supervisor who is not involved in the evaluation of outcome parameters to ensure blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Relaxation intervention with natural sounds (Experimental): The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with nature sounds.
  Interventions: Device: Intervention with natural sounds administered via headphones
- Relaxation intervention with natural sounds and binaural beats (Experimental): The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with nature sounds and binaural beats.
  Interventions: Device: Intervention with natural sounds and binaural beats administered via headphones
- Relaxation intervention with natural sounds and virtual reality (Experimental): The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with a nature scene in a spherical 360° environment with associated nature sounds.
  Interventions: Device: Intervention with natural sounds and virtual reality administered via headphones and head mounted display
- Relaxation intervention with natural sounds, binaural beats and virtual reality (Experimental): The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with a nature scene in a spherical 360° environment with associated nature sounds and binaural beats.
  Interventions: Device: Intervention with natural sounds, binaural beats and virtual reality administered via headphones and head mounted display
- Control without Intervention (No Intervention)

INTERVENTIONS:
Device: Intervention with natural sounds administered via headphones — The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with nature sounds.
  Arms: Relaxation intervention with natural sounds
Device: Intervention with natural sounds and binaural beats administered via headphones — The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with nature sounds and binaural beats.
  Arms: Relaxation intervention with natural sounds and binaural beats
Device: Intervention with natural sounds and virtual reality administered via headphones and head mounted display — The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with a nature scene in a spherical 360° environment with associated nature sounds.
  Arms: Relaxation intervention with natural sounds and virtual reality
Device: Intervention with natural sounds, binaural beats and virtual reality administered via headphones and head mounted display — The preoperative intervention includes a stress-reducing relaxation phase lasting approximately 30 minutes, during which the patients are presented with a nature scene in a spherical 360° environment with associated nature sounds and binaural beats.
  Arms: Relaxation intervention with natural sounds, binaural beats and virtual reality

SUMMARY:
Patients undergoing cardiac surgery often complain of anxiety before a major operation and the resulting stress. This circumstance is a risk factor for mental problems that may occur after the operation (e.g., delirium or memory deficits). This study aims to prevent these discomforts by a preoperative relaxation intervention.

DETAILED DESCRIPTION:
Preoperative anxiety and stress are risk factors for postoperative delirium (PD), postoperative cognitive decline (POCD), morbidity, and mortality. The primary objective of this study is to reduce the preoperative stress response through the combined presentation of a virtual reality environment with natural landscape and binaural beats. The proposed study is a monocenter, 5-arm prospective randomized controlled intervention of 125 patients undergoing elective cardiac surgery using extracorporeal circulation. A 360 ° video sequence including natural sounds (with and without binaural beats) are presented to 2 groups, and 2 groups receive only natural sounds (with and without binaural beats); a group without stimuli (standard procedure) represents the control group.

On the day of admission to the acute care clinic, a detailed examination of neuropsychological functions and health-related quality of life (HQL) is scheduled. Cortisol-saliva, heart rate variability and electrodermal activity as indicators for stress and relaxation are measured during the intervention phase (duration: approximately 30 minutes), which leads directly into the narcosis phase.

To investigate postoperative neurocognitive dysfunctions, daily delirium screenings will be performed after surgery, and a neuropsychological examination will be performed at the time of discharge from the acute hospital and at 3 months after surgery. Changes in HQL will also be completed at 3 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elective cardiac surgery (coronary artery bypass surgery, aortic or mitral valve replacement/reconstruction, or combination surgery) with standardized extracorporeal circulation.
2. A sufficiently good knowledge of German is necessary as neuropsychological tests are language-dependent.

Exclusion Criteria:

1. History of acute clinically relevant cognitive impairment of any cause (e.g., dementia, depression, stroke, multiple sclerosis) that may impair neuropsychological evaluation.
2. Contraindications to the presentation of binaural beats or visual stimuli (e.g., epilepsy),
3. Significant hearing loss or astigmatism, which may interfere with optimal perception of auditory and visual stimuli.
4. Taking sedatives on the day of surgery.
5. Unwilling to participate in the relaxation procedure or neuropsychological testing due to deteriorating health, lack of motivation, or other reasons.
6. Participation in interventions that aim to change cognitive or emotional functioning which cannot be systematically controlled by our study team.
7. Participation in an interventional study according to AMG/MPG will also be excluded.
8. Patients with missing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-RMSSD | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-NN50 | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-pNN50 | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-HF | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-HF% | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-VLF | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-VLF% | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-LF | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-LF% | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-LF/HF | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-SD1 | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline heart rate variability (HRV) at the end of intervention as assessed using ECG-SD2 | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention

SECONDARY OUTCOMES:
Change from baseline cortisol at the end of intervention as assessed using saliva | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline oxytocin at the end of intervention as assessed using saliva | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline alpha-amylase at the end of intervention as assessed using saliva | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline cortisol at the end of intervention as assessed using blood sample | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline oxytocin at the end of intervention as assessed using blood sample | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline alpha-amylase at the end of intervention as assessed using blood sample | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline electro dermal activity (EDA) at the end of intervention as assessed using EDA-SCL | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline electro dermal activity (EDA) at the end of intervention as assessed using EDA-NS-SCRs | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Change from baseline bispectral index (BIS) at the end of intervention | Approximately 30 minutes. Immediately pre-intervention to Immediately post-intervention
Amount of propofol during induction of narcosis | Immediately pre-induction of narcosis to immediately post-induction of narcosis
Amount of sufentanil during induction of narcosis | Immediately pre-induction of narcosis to immediately post-induction of narcosis
Amount of remifentanil during induction of narcosis | Immediately pre-induction of narcosis to immediately post-induction of narcosis
Amount of propofol during surgery phase | Immediately post-induction of narcosis to immediately post-narcosis
Amount of sufentanil during surgery phase | Immediately post-induction of narcosis to immediately post-narcosis
Amount of remifentanil during surgery phase | Immediately post-induction of narcosis to immediately post-narcosis
Duration of stay at intensive care unit | Immediately post-surgery to approximately 1-2 days post-surgery
Duration of stay at normal ward | Immediately post-intensive care unit to approximately 1 week post-intensive care unit
Number of participants with postoperative delirium during the stay in the intensive care unit as assessed using the "Intensive Care Delirium Screening Checklist" (ICDSC) | Immediately post-surgery to approximately 1-2 days post-surgery
  Postoperative delirium is defined as the occurrence of at least one delirious episode during a stay in the intensive care unit. The "Intensive Care Delirium Screening Checklist" (ICDSC) records the clinical symptoms of consciousness, attention, orientation, hallucinations, psychomotor retardation or agitation and speech.
Number of participants with postoperative delirium during the stay on normal ward as assessed using the "Confusion Assessment Method" (3D-CAM) | Immediately post-intensive care unit to approximately 1 week post-intensive care unit
  Postoperative delirium is defined as the occurrence of at least one delirious episode during a stay in an intensive care unit or normal ward. The "Confusion Assessment Method" (3D-CAM) records the clinical symptoms of consciousness, attention, orientation, hallucinations, psychomotor retardation or agitation and speech.
Number of participants with postoperative cognitive decline at the time of discharge from the acute clinic, defined as a decrease between the pre- and postoperative examinations of one standard deviation measured with the "Montreal Cognitive Assessment" | Approximately 1 day pre-surgery to approximately 9 days post-surgery
  The "Montreal Cognitive Assessment" (MOCA) is a screening procedure for general cognitive function.
Number of participants with postoperative cognitive decline at 3 months after surgery, defined as a decrease between pre- and postoperative examinations of one standard deviation in at least 20% of all objective neuropsychological parameters | Approximately 1 day pre-surgery to 3 months post-surgery
  The objective neuropsychological parameters measure cognitive domains such as immediate memory span, free recall, recognition memory, selective attention, working memory, word fluency, inhibition, spatial imagination, visuoconstructive ability, and recognition of emotions. These cognitive domains will be measured with the following instruments: "Verbal Learning and Memory Test (VLMT), "Brief Visuospatial Memory Test-Revised" (BVMT-R), "Trail Making Test A/B" (TMT), "Letter Number Span Test" (LNS), "Regensburger Wordfluency-Test" (RWT), "Syndrom-Short Test/Inhibition" (in german: Syndrom-Kurz Test, SKT-7), "Performance Testing System" (in german: "Leistungsprüfsystem", LPS-9), "3-D Figure/Montreal Cognitive Assessment" (MOCA-3-D-Figure), and "Penn Emotion Recognition Test" (ER40).
Number of participants with subjective postoperative cognitive decline (POCD-S) at 3 months after surgery, defined as a subjective decrease between pre- and postoperative examinations of one cognitive function. | Immediately post-surgery to 3 months post-surgery
  The "Subjective Postoperative Cognitive Decline" (POCD-S) questionnaire assesses the occurrence of postoperative cognitive deficits (memory, attention, executive functions, language, and orientation) that appeared specifically as a result of the cardiac surgery.
Number of participants with deficits in instrumental activity of daily living (IADL) at 3 months after surgery, defined as the occurrence of at least one deficit. | Immediately post-surgery to 3 months post-surgery
  The "Instrumental Activity of Daily Living" (IADL) questionnaire assesses the occurrence of deficits in the domains of cooking, telephoning, shopping, light and heavy housework, and organizing (finances, taking medications).
Change from baseline visual immediate memory span at 3 months post-surgery as assessed using the "Brief Visuospatial Memory Test-Revised" (BVMT-R) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Brief Visuospatial Memory Test-Revised" (BVMT-R), the patient is shown six geometric figures for 10 seconds on a DIN A4 sheet of paper, which are to be drawn directly afterward. This procedure is repeated with the same figures in a total of three learning trials. The figures are to be freely replicated in a time-delayed episode with following recognition help.
Change from baseline visual free recall at 3 months post-surgery as assessed using the "Brief Visuospatial Memory Test-Revised" (BVMT-R) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Brief Visuospatial Memory Test-Revised" (BVMT-R), the patient is shown six geometric figures for 10 seconds on a DIN A4 sheet of paper, which are to be drawn directly afterward. This procedure is repeated with the same figures in a total of three learning trials. The figures are to be freely replicated in a time-delayed episode with following recognition help.
Change from baseline visual recognition memory at 3 months post-surgery as assessed using the "Brief Visuospatial Memory Test-Revised" (BVMT-R) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Brief Visuospatial Memory Test-Revised" (BVMT-R), the patient is shown six geometric figures for 10 seconds on a DIN A4 sheet of paper, which are to be drawn directly afterward. This procedure is repeated with the same figures in a total of three learning trials. The figures are to be freely replicated in a time-delayed episode with following recognition help.
Change from baseline verbal immediate memory span at 3 months post-surgery as assessed using the "Verbal Learning and Memory Test" (VLMT) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Verbal Learning and Memory Test" (VLMT), a list of words is learned over five learning trials. After an interference word list, the initial word list is to be remembered directly and with a delay of about 20 minutes. With subsequent recognition help, the verbal discrimination ability is measured.
Change from baseline verbal free recall at 3 months post-surgery as assessed using the "Verbal Learning and Memory Test" (VLMT) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Verbal Learning and Memory Test" (VLMT), a list of words is learned over five learning trials. After an interference word list, the initial word list is to be remembered directly and with a delay of about 20 minutes. With subsequent recognition help, the verbal discrimination ability is measured.
Change from baseline verbal recognition memory at 3 months post-surgery as assessed using the "Verbal Learning and Memory Test" (VLMT) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Verbal Learning and Memory Test" (VLMT), a list of words is learned over five learning trials. After an interference word list, the initial word list is to be remembered directly and with a delay of about 20 minutes. With subsequent recognition help, the verbal discrimination ability is measured.
Change from baseline selective attention at 3 months post-surgery as assessed using the "Trail Making Test A" (TMT-A) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Trail Making Test A" (TMT-A), the patient has to connect numbers in ascending order on a test sheet as fast as possible.
Change from baseline verbal working memory at 3 months post-surgery as assessed using the "Letter Number Span Test" (LNS) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Letter Number Span Test" (LNS), the patient is supposed to rearrange a mixed sequence of letters and numbers through mental reorganization in such a way that first all numbers and then all letters are to be named in ascending order.
Change from baseline cognitive flexibility at 3 months post-surgery as assessed using the "Trail Making Test B" (TMT-B) | Approximately 1 day pre-surgery to 3 months post-surgery
  With the "Trail Making Test B" (TMT-B), the patient's task is to connect numbers and letters alternately in ascending order.
Change from baseline inhibition at 3 months post-surgery as assessed using the "Syndrom-Short Test/Inhibition" (in german: Syndrom-Kurz Test, SKT-7) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Syndrom-Short Test/Inhibition" (in german: Syndrom-Kurz Test, SKT-7), the patient has to rename a series of letters (e.g., "A" instead of "B," and vice versa).
Change from baseline category word fluency at 3 months post-surgery as assessed using the "Regensburger Wordfluency-Test" (RWT) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Regensburger Wordfluency-Test" (RWT), the patient has to name in 1 minute as many words as possible from a certain category.
Change from baseline phonetic word fluency at 3 months post-surgery as assessed using the "Regensburger Wordfluency-Test" (RWT) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Regensburger Wordfluency-Test" (RWT), the patient has to name in 1 minute as many words as possible with a certain initial letter.
Change from baseline spatial imagination at 3 months post-surgery as assessed using the "Performance Testing System" (in german: "Leistungsprüfsystem", LPS-9) | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Performance Testing System" (in german: "Leistungsprüfsystem", LPS-9), the patient has to count in 3 minutes as many surfaces of a 3-D geometric figure as possible.
Change from baseline visuoconstructive ability at 3 months post-surgery as assessed using the subtest "3-D figure copy" of the "Montreal Cognitive Assessment" (MOCA). | Approximately 1 day pre-surgery to 3 months post-surgery
  In the subtest "3-D figure copy" of the "Montreal Cognitive Assessment" (MOCA), the patient has to copy a 3 dimensional geometric figure.
Change from baseline recognition of emotions at 3 months post-surgery as assessed using the "Penn Emotion Recognition Test" (ER40). | Approximately 1 day pre-surgery to 3 months post-surgery
  In the "Penn Emotion Recognition Test" (ER40), the patient has to select the correct emotion label (joy, sadness, anger, fear, and neutral) for each facial expression.
Change from baseline cognitive failures in everyday life at 3 months after surgery as assessed using the "Cognitive Failures Questionnaire" (CFQ) | Approximately 1 day pre-surgery to 3 months post-surgery
  The "Cognitive Failures Questionnaire" (CFQ) measures the frequency of failures in daily living in terms of memory, attention, action, and perception.
Change from baseline health-related quality of life at 3 months after surgery as assessed using the "36-Item Short Form Health Survey" (SF36) | Approximately 1 day pre-surgery to 3 months post-surgery
  The "36-Item Short Form Health Survey" (SF36) includes 36 questions covering 8 health-related factors: vitality, physical functioning, bodily pain, general health perception, physical role function, emotional role function, social role functioning, and mental health.
Change from baseline depression at 3 months after surgery as assessed using the subscale "Depression" of the "Hospital Anxiety and Depression Scale" (HDS) | Approximately 1 day pre-surgery to 3 months post-surgery
  The subscale "Depression" of the "Hospital Anxiety and Depression Scale" (HDS) includes 7 questions covering core features of typical depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kerckhoff Heart Center, Heart and Brain Research Group, Bad Nauheim, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified participants' data analyzed during the current study will be available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Up to one year after publication of the data
Access Criteria: IPD will be available on reasonable request.